CLINICAL TRIAL: NCT01508728
Title: Efficacy Study of a Sensory Feedback Knee Orthosis in Patients Suffering From Unoperated Severe Knee Sprain
Acronym: ORTHOSENS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011-A00821-40; 2011-A00821-40 (Other: AFSSAPS (N° ID RCB))
Record Dates: First submitted 2012-01-03; First posted 2012-01-12 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Sprain
Keywords: unoperated severe sprain of the knee with partial or total rupture of the anterior; cruciate ligament and medial or lateral collateral ligament
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Active vibration (Experimental)
  Interventions: Device: ORTHOSENS orthosis
- Placebo Vibration (Placebo Comparator)
  Interventions: Device: ORTHOSENS orthosis

INTERVENTIONS:
Device: ORTHOSENS orthosis — with active vibration
  Arms: Active vibration
Device: ORTHOSENS orthosis — with placebo vibration
  Arms: Placebo Vibration

SUMMARY:
Ortheses are commonly used for the repair of damage to the musculoskeletal system. However, immobility, by itself, causes serious side effects that require long and costly rehabilitation. The Sensory Feedback Ortheses allow to artificially maintain the proprioceptive and tactile flow in order to maintain the activity of their host brain areas and thus reduce significantly the usual therapy duration. The clinical study Orthosens will evaluate the efficacy and safety of the Sensory Feedback Ortheses.

ELIGIBILITY:
Inclusion Criteria:

* Patients agreeing to participate in the study and who signed informed consent.
* Indication of bracing immobilization for 6 weeks following a unoperated severe sprain of the knee with partial or total rupture of the anterior cruciate ligament and a peripheral injury, medial or lateral collateral ligament, with or without meniscal lesion.
* MRI scan confirming the nature of the lesion to be provided

during the inclusion visit.

* Patients whose knee is immobilized for 7 to 15 days in Zimmer-like splint.
* Patients aged from 18 to 65.
* Patients agreeing to choose their physiotherapist from a list provided by the investigators.
* Patient (s) with insurance coverage.

Exclusion Criteria:

* Patients with a bucket handle meniscus tear.
* Patients with a pentad injury.
* Patients with osteochondral fragments.
* Patients with a knee fracture apart from "Segond fracture" and "bone bruise".
* Patients who underwent ligament surgery for the concerned knee.
* Patients with a bone lesion which may interfere with the knee joint(distal femur, proximal tibia, patella).
* Patients with any history of rupture of the central pivot (anterior cruciate ligament and posterior cruciate ligament), of lateral ligament planes rupture (medial collateral ligament and lateral collateral) or lateral planes ligament injury without rupture, dating from less than 1 year.
* Patients whose sprain results from an accident at work.
* Patients with an inability / unwillingness to follow protocol requirements.
* Patients for whom there would be no suitable brace size in the Thuasne range.
* Patients participating in another clinical study or who have tested an experimental drug within 30 days prior to study entry. - Patients with another disease which, according to the investigator, may interfere with the results or the conduct of the trial and thus justify their non-inclusion in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Period of time required to recover a normal knee range of motion

SECONDARY OUTCOMES:
Period of time required to recover a normal knee range of motion with a passive mobilization | The day of inclusion, then 3 times per week during 12 weeks (except at weeks 8 and 12: 4 measurements)
Pain according to Visual Analogic Scale | The day of inclusion, then 3 times per week during 12 weeks (except at weeks 8 and 12: 4 measurements)
Safety according to adverse event records | At any time during subject participation (12 weeks)
Psychological state according to the Incredibly Short Profile of Mood States | 3 times per week from week 1 to week 12
Knee functional state according to IKDC, KOOS and KOOS-PS scores | The Day of inclusion, then 3 times per week during 12 weeks (except at weeks 8 and 12: 4 measurements)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Clinique Axium, Aix-en-Provence
  - Institut de Chirurgie Orthopédique et Sportive, Marseille
  - Hôpital Sainte-Marguerite, Marseille